CLINICAL TRIAL: NCT02763553
Title: Does a Ketogenic Diet Reduce Delirium in Intensive Care? Part 1: - A Feasibility Study to Test if a Ketogenic Diet Causes Ketosis in Patients on Intensive Care
Brief Title: Does a Ketogenic Diet Causes Ketosis in Patients on Intensive Care?
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospitals Bristol and Weston NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN/2015/5042
Record Dates: First submitted 2016-04-26; First posted 2016-05-05 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Ketosis
Keywords: Ketone Bodies; Enteral Nutrition; Ketogenic Diet
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketogenic Feed (Experimental): A low-carbohydrate, high-fat enteral feed (Nutrison KetoCal 4:1) containing 0.4g of carbohydrate and 10g of fat per 100kcal. Given as a continuous feed via a naso-gastric tube as per standard feeding protocol.
  Interventions: Dietary Supplement: Ketogenic Feed
- Standard Feed (Active Comparator): Standard enteral feed (Nutrison ProteinPlus MF 1.28) containing 11.1g of carbohydrate and 3.8g of fat per 100kcal. Given as a continuous feed via a naso-gastric tube as per standard feeding protocol.
  Interventions: Dietary Supplement: Standard Feed

INTERVENTIONS:
Dietary Supplement: Ketogenic Feed — A low-carbohydrate, high-fat feed designed to induce a ketotic state.
  Other Names: Nutrison KetoCal 4:1
  Arms: Ketogenic Feed
Dietary Supplement: Standard Feed — Standard enteral feed used in critical care patients requiring nutrition via a nasogastric tube
  Other Names: Nutrison ProteinPlus MultiFibre 1.28
  Arms: Standard Feed

SUMMARY:
The purpose of this study is to assess if an enteral ketogenic feed will cause a ketotic state in critically ill patients on intensive care.

DETAILED DESCRIPTION:
This pilot study is a prospective, single-centre, unblinded, parallel-group, randomised controlled, Phase IIb trial comparing standard enteral nutrition with an enteral ketogenic feed. The trial has a simple, pragmatic design and will be analysed on an intention-to-treat basis. It aims to recruit 10 patients from a single University teaching hospital adult general ICU. The anticipated recruitment period is 4 weeks.

Adult patients admitted to intensive care and expected to require enteral feed via a nasogastric tube for at least 5 days and who fulfil other eligibility criteria will be allocated at random to receive either standard feed (Nutrison Protein Plus Multi Fibre) or a ketogenic enteral feed (Nutrison KetoCal 4:1).

The primary endpoint will be increase in ketone body concentration in serum. Secondary endpoints will include, time taken to achieve a ketotic state, ketone levels in critical care patients who are not absorbing enteral feed, glucose levels in patients on a ketone feed, triglyceride and cholesterol levels, creatinine kinase levels and development of a metabolic acidosis.

Adult ICU patients will be eligible to be included in this study if they are expected to require enteral feed via a nasogastric or nasojejunal tube or established percutaneous jejunostomy for at least 5 days. Practically, this will be achieved by screening ventilated patients as they will require enteral feeding Major exclusion criteria include contraindications to ketogenic feeds, contraindications to enteral feeding, a new (< 5 days) percutaneous jejunostomy.

The intervention will continue until 14 days if the patient still requires enteral nutrition or until able to commence a normal diet orally.

ELIGIBILITY:
Inclusion Criteria:

* Adults who require mechanical ventilation within 72 hours of admission to intensive care

Exclusion Criteria:

* Known intolerance to the ketogenic diet
* Contraindication to standard protocolised enteral feeding
* Pregnancy
* Severe liver disease (known decompensated liver cirrhosis, previous liver transplant, acute hepatitis (bilirubin >100, ALT >500)
* Severe metabolic acidosis (pH < 7.2, HCO3 < 15mmol/L) that has not been corrected prior to enrolment in the study
* Patients predicted to stay less than 24 hours on intensive care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-01 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Median serum ketone level | 14 days
  Serum ketone levels (mmol/L) will be recorded 4-hourly in each group. The median serum ketone level (mmol/L) will be calculated.

SECONDARY OUTCOMES:
Time to achieve serum ketosis | 14 days
  Time taken (hours) to achieve a clinically relevant ketosis (serum ketone > 0.3mmol/L) from introduction of an enteral ketogenic feed.

CONTACTS AND LOCATIONS:
Overall Officials: Kieron D Rooney, MBBS, Study Chair — University Hospitals Bristol and Weston NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: Yes
No, anonymised data only